CLINICAL TRIAL: NCT02736981
Title: Low Intensity Weight Loss for Young Adults
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20002772; R01DK103668 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-04-13 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Young Adults
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral Weight Loss (BWL) (Active Comparator): 24 week treatment program consisting of a single, 90-minute, in-person group session in week 1, and a single 45 minute individual in-person session in week two, followed by a 6 month technology mediated program. The program includes evidenced-based behavioral weight loss content, individualized diet and physical activity goals, weekly lessons as well as reporting of key behaviors and personalized feedback to aid in goal attainment.
  Interventions: Behavioral: Behavioral Weight Loss (BWL)
- BWL + Autonomous Motivation (Active Comparator): 24 week treatment program consisting of a single, 90-minute, in-person group session in week 1, and a single 45 minute individual in-person session in week two, followed by a 6 month technology mediated program. The program includes evidenced-based behavioral weight loss content, individualized diet and physical activity goals, weekly lessons as well as reporting of key behaviors and personalized feedback to aid in goal attainment. Participants in this arm will receive coaching that places an increased emphasis on their values and personal choices, and also have the option to attend several experiential group sessions that will help those interested to apply the material and skills they are being taught (e.g., cooking demonstration, circuit training class).
  Interventions: Behavioral: Behavioral Weight Loss (BWL); Behavioral: BWL + Autonomous Motivation
- BWL + Extrinsic Motivation (Active Comparator): 24 week treatment program consisting of a single, 90-minute, in-person group session in week 1, and a single 45 minute individual in-person session in week two, followed by a 6 month technology mediated program. The program includes evidenced-based behavioral weight loss content, individualized diet and physical activity goals, weekly lessons as well as reporting of key behaviors and personalized feedback to aid in goal attainment. Participants in this arm will have the opportunity to receive small monetary incentives in weeks 2-24 for tracking weight and calorie intake, and will be eligible for a raffle based on weight loss.
  Interventions: Behavioral: Behavioral Weight Loss (BWL); Behavioral: BWL + Extrinsic Motivation

INTERVENTIONS:
Behavioral: Behavioral Weight Loss (BWL) — The intervention represents an adapted version of gold-standard evidence based adult behavioral weight loss that has been tailored specifically to meet the needs of 18-25 year olds. The program includes personalized dietary and physical activity prescriptions, training in behavioral strategies, weekly lesson content, and reporting of key behaviors and personalized feedback and coaching.
Behavioral: BWL + Autonomous Motivation — The intervention represents an adapted version of gold-standard evidence based adult behavioral weight loss that has been tailored specifically to meet the needs of 18-25 year olds. The program includes personalized dietary and physical activity prescriptions, training in behavioral strategies, weekly lesson content, and reporting of key behaviors and personalized feedback and coaching. Participants in this arm will receive coaching that places an increased emphasis on their values and personal choices, and also have the option to attend several experiential group sessions that will help those interested to apply the material and skills they are being taught (e.g., cooking demonstration, circuit training class).
  Arms: BWL + Autonomous Motivation
Behavioral: BWL + Extrinsic Motivation — The intervention represents an adapted version of gold-standard evidence based adult behavioral weight loss that has been tailored specifically to meet the needs of 18-25 year olds. The program includes personalized dietary and physical activity prescriptions, training in behavioral strategies, weekly lesson content, and reporting of key behaviors and personalized feedback and coaching. Participants in this arm will have the opportunity to receive small monetary incentives in weeks 2-24 for tracking weight and calorie intake, and will be eligible for a raffle based on weight loss.
  Arms: BWL + Extrinsic Motivation

SUMMARY:
This is a 3-arm randomized controlled trial to test the efficacy of three novel motivational approaches to weight loss with 18-25 year olds. Participants will be 18-25 year olds with a BMI of 25-45 kg/m2, randomized to: 1) Behavioral Weight Loss (BWL), 2) BWL + Autonomous Motivation (BWL+Aut) or 3) BWL + Extrinsic Motivation (BWL+Ext). All arms will receive a 6-month behavioral weight loss intervention, followed by a 6-month no-treatment follow up period.

DETAILED DESCRIPTION:
A 3-arm randomized controlled trial will be conducted, the goal of which is to determine which group represents the most viable approach to behavioral weight loss treatment with 18-25 year olds. A total of 381 participants,18-25 years of age, with a BMI between 25 and 45 kg/m2 will be randomized to one of three groups: 1) Behavioral Weight Loss (BWL), 2) BWL + Autonomous Motivation (BWL+Aut) or 3) BWL + Extrinsic Motivation (BWL+Ext). All arms will receive a 24-week behavioral weight loss intervention, including personalized dietary, physical activity, and weight loss prescriptions. In addition, all arms will be followed for a 6 month no treatment follow-up period. Assessments of weight and secondary outcomes will occur in 0, 3, 6 and 12 months. The investigators will compare treatment effects, across all 3 arms at 6 months, and compare arms on weight loss maintenance at12 months. The investigators will also examine mediators of treatment outcomes consistent with the investigators theoretical framework.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-25 years of age. Body Mass Index (BMI) between 25 and 45 kg/m2. Men and women will be recruited. All race and ethnic groups will be recruited.

Exclusion Criteria:

* Report an uncontrolled medical condition that may pose a safety issue given the recommendations for diet and unsupervised physical activity in the current study (e.g., uncontrolled hypertension). The investigators will refer individuals who have blood pressure levels >140 / 90 mmHg as part of baseline screening to their physician and exclude them from this study unless their treating physician determines s/he is a suitable candidate based on the specifics of the protocol and provides written medical consent for participation. Participants who report a history of or current treatment for medical conditions (e.g., hypertension, diabetes) will be asked to obtain MD consent to participate.
* Other health problems or medications which may influence the ability to walk for physical activity or be associated with unintentional weight change, including cancer treatment within the past 5 years or tuberculosis.
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q), which will be administered during prescreen. Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
* Report a history of, or current diagnosis of anorexia nervosa or bulimia nervosa, or any current compensatory behaviors (e.g., vomiting, laxative use, excessive exercise).
* Current symptoms of alcohol or substance dependence.
* Planning to move from the area within the study period.
* Currently pregnant, pregnant within the past 6 months, currently breastfeeding or planning to become pregnant within the next 12 months.
* Hospitalization for depression or other psychiatric disorder within the past 12 months. History of psychotic disorder or bipolar disorder.
* Another member of the household is a participant or staff member on this study.
* Participation in another research study that may interfere with this study.
* Currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 3 months.
* Failure to complete the screening appointments.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 382 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2020-02-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 6 Months
  Primary pre-specified outcome is weight change in kilograms from baseline to 6 months. Change in kg was used in power calculations.
Percent Weight Loss | 6 Months
  Pre-specified analyses to examine impact on weight include percent weight loss from baseline to 6 months
Change in Body Mass Index | 6 Months
  Change in body mass index (calculated as change in kg/m^2, weight in kilograms, height in meters) from baseline to 6 months.

SECONDARY OUTCOMES:
Waist Circumference | 6 Months
  Change in waist circumference (in cm) from baseline to 6 months.
Body Composition (percent fat mass) | 6 Months
  Change in fat mass from baseline to 6 months, measured by bioelectrical impedance analysis.
Blood Pressure | 6 Months
  Change in systolic blood pressure (SBP) and diastolic blood pressure (DBP) from baseline to 6 months.
Minutes of Moderate to Vigorous Physical Activity | 6 Months
  Change in minutes of moderate-to-vigorous activity from baseline to 6 months as assessed by objective activity monitors (Actigraph).
Dietary Intake | 6 Months
  Change in fat intake, sugared beverage intake, alcohol intake, fruit and vegetable intake from baseline to 6 months as assessed by interviewer administered modules.

OTHER OUTCOMES:
Weight Loss Maintenance | 12 Months
  Pre-specified analyses to examine overall weight loss maintenance include weight change in kilograms from baseline to 12 months and change in percent weight loss from baseline to 12 months. Please note that both indices were included in the same secondary aim for funding agency and approved.
Long-term Change in Body Mass Index | 12 Months
  Overall change in body mass index (calculated as change in kg/m^2) from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, School of Medicine, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LaRose JG, Leahey TM, Lanoye A, Bean MK, Fava JL, Tate DF, Evans RK, Wickham EP 3rd, Henderson MM. Effect of a Lifestyle Intervention on Cardiometabolic Health Among Emerging Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231903. doi: 10.1001/jamanetworkopen.2022.31903. PMID 36121656
- [Derived] LaRose JG, Leahey TM, Lanoye A, Bean MK, Tate DF, Fava JL, Evans RK, Wickham E 3rd, Henderson MM, Hatley K, Diamond M. Behavioral weight loss in emerging adults: Design and rationale for the Richmond Emerging Adults Choosing Health (REACH) randomized clinical trial. Contemp Clin Trials. 2021 Aug;107:106426. doi: 10.1016/j.cct.2021.106426. Epub 2021 May 24. PMID 34044124
- [Derived] Brown KL, Hines AL, Hagiwara N, Utsey S, Perera RA, LaRose JG. The Weight of Racial Discrimination: Examining the Association Between Racial Discrimination and Change in Adiposity Among Emerging Adult Women Enrolled in a Behavioral Weight Loss Program. J Racial Ethn Health Disparities. 2022 Jun;9(3):909-920. doi: 10.1007/s40615-021-01030-7. Epub 2021 Mar 29. PMID 33782906

DOCUMENTS (1):
  • Informed Consent Form (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02736981/ICF_000.pdf